CLINICAL TRIAL: NCT04554004
Title: A Clinical Trial for CT Myocardial Perfusion Based Non-invasive Index of Microciculatory Resistance
Brief Title: A Non-invasive Index of Microciculatory Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jinyu Huang, professor, First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020C03018
Record Dates: First submitted 2020-09-08; First posted 2020-09-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Coronary Microvascular Disease; Coronary Artery Disease
MeSH Terms: conditions — Microvascular Angina; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All consecutive patients undergoing outine CT angiography and dynamic CT-myocardial perfusion imaging(MPI) will be potentially eligible for inclusion in the trial. Assessment of coronary stenosis severity using invasive fractional flow reserve (FFR) and the status of myocardial microcirculation perfusion including coronary flow reserve (CFR) and index of microvascular resistance (IMR) will be performed as part of invasive coronary angiography(CAG).
  Interventions: Diagnostic Test: CCTA, CT-MPI, DSA, FFR

INTERVENTIONS:
Diagnostic Test: CCTA, CT-MPI, DSA, FFR — The patients who enrolled the study will undergo coronary CT angiography(CCTA), dynamic CT-MPI, invasive coronary angiography and invasive computation of fractional flow reserve (FFR)

SUMMARY:
Coronary artery microvascular disease (CMVD) lacks reliable and non-invasive quantitative diagnosis methods. Improving coronary microcirculation has become one of the main goals of coronary heart disease treatment. In this study, by establishing the key influencing factors of myocardial microcirculation perfusion, an accurate three-dimensional reconstruction method of coronary artery was established, and a non-invasive coronary microcirculation resistance index (CT-IMR) calculation method based on computational fluid method mechanics was established. At the same time, a phase I single-center clinical verification and a multi-center clinical verification of the non-invasive coronary microcirculation function precision assessment system were carried out, and a non-invasive coronary microcirculation detection system and technology were established.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be older than 18 years
* Written informed consent available
* Subject is indicated for invasive coronary angiography
* Subject need to be taken within 30 days after enrolment

Exclusion Criteria:

* Previous PCI or CABG
* Subject is not eligible for measuring IMR
* Complicated complex congenital heart disease
* Artificial pacemaker or internal defibrillator leads implanted
* Implanted artificial heart valve
* Severe arrhythmia including complete AV block, ventricular arrhythmia
* Impaired chronic renal function (serum creatinine>1.5ULN)
* Allergic to iodine
* Pregnancy
* Body mass index >35 kg/m2
* Left ventricle is markedly thickened
* Needs for emergency procedures
* Severe distortion of in the blood vessel
* Unstable haemodynamics including abrupt chest pain cardiogenic shock, unstable blood pressure (systolic < 90mmHg), severe congestive heart failure or pulmonary edema
* Life-threatening diseases (life expectancy < 2 months)
* Tako Tsubo syndrome (TTS)
* Others who are inappropriate subject judged by clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity | up to 12 months
  The sensitivity and specificity of CT-IMR in the diagnosis of microcirculation dysfunction were studied.

SECONDARY OUTCOMES:
diagnostic | up to 12 months
  To study the diagnostic coincidence rate, positive predictive value and negative predictive value of CT-IMR in the diagnosis of microcirculation dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- First People's Hospital of Hangzhou, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (text, table, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: When will data be available (start and end dates)?Beginning 3 months. No end data.
Access Criteria: Proposals should be directed to zdsyhjy0902@zju.edu.cn. To gain access, data requestors will need to sign a data access agreement.